CLINICAL TRIAL: NCT04020406
Title: In Vitro Evaluation of Antibacterial Activity of Urea Solution Against Ocular Bacterial Isolates
Brief Title: Antibacterial Activity of Urea Against Ocular Bacteria
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Lotfy Fahmy, Clinical Professor, Assiut University
Other Study IDs: 2323297
Record Dates: First submitted 2019-07-07; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Urea in Blood; High
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Antibacterial Activity of Urea: Activity of Urea Solution against Ocular Bacterial Isolates
  Interventions: Biological: Antibacterial Activity

INTERVENTIONS:
Biological: Antibacterial Activity — Antibacterial Activity of Urea Solution against Ocular Bacterial Isolates

SUMMARY:
Antibacterial properties of urea was tested against 35 isolates from ocular infections.

DETAILED DESCRIPTION:
In vitro susceptibility testing was performed with commercially available antibiotic discs, homemade urea discs saturated with urea solution at a concentration of 96 mmol. The weight of urea in one drop = 0.37 mg, in one ml = 10.34 mg (5 microliter/ disc) discs and combined discs (antibiotic discs to which urea solution was added). Combined discs provided better in vitro susceptibility results than antibiotics alone.

Scanning electron micrographs of bacterial isolates incubated overnight with urea solution showed marked disruption of bacterial aggregative patterns and irregularities of their cell walls.

Western blotting showed marked reduction in total proteins in bacterial isolates incubated overnight with urea solution. These findings may explain the possible mechanisms for antibacterial activity of urea solution as a result of protein denaturation.

ELIGIBILITY:
Inclusion Criteria:

* ocular infection

Exclusion Criteria:

* Local antibiotics treatment

Ages: 5 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: individuals with any ocular infection
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Antibacterial effect of Urea Solution against Ocular Bacterial | 6 month
  Samples were both inoculated on Muller Agar (Sigma-Aldrich) plates and directly examined under the microscope using Gram stained smears. Inoculated plates were incubated at 37oC for 48 hrs.
  Gram negative isolates were sub-cultured on MacConkey's, Eosin Methelyene Blue (EMB) and Cystine Lactose Electrolyte Deficient (CLED) agar plates (Sigma-Aldrich). Gram positive isolates were sub-cultured on Mannitol Salt agar plates (Sigma-Aldrich).

CONTACTS AND LOCATIONS:
Overall Officials: Hassan 58 Lotfy, Professor, Principal Investigator — Assiut T
Locations (1):
- Hassan Lotfy Fahmy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided